CLINICAL TRIAL: NCT06221748
Title: A Randomized，Multicenter, Open-Label，Phase II/III Study to Evaluate the Safety and Efficacy of Disitamab Vedotin Combined With Cadonilimab in Subjects With HER2-expressing Locally Advanced or Metastatic Gastric Cancer and Gastroesophageal Junction Adenocarcinoma Who Have Progressed on r First-line Therapy
Brief Title: DV Combined With Cadonilimab in Subjects With HER2-expressing Gastric Cancer and Gastroesophageal Junction Adenocarcinoma After Progression on First-line Therapy
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: RemeGen Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RC48-C035
Record Dates: First submitted 2024-01-15; First posted 2024-01-24 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2024-01

CONDITIONS: Gastric Cancer; Gastroesophageal Junction Adenocarcinoma
Keywords: Gastric cancer; Gastroesophageal junction adenocarcinoma; HER2- expressing
MeSH Terms: conditions — Stomach Neoplasms | interventions — disitamab vedotin; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Disitamab Vedotin + Cadonilimab (Experimental): Disitamab Vedotin With Cadonilimab
  Interventions: Drug: Disitamab Vedotin Injection; Drug: Cadonilimab Injection
- Disitamab Vedotin (Experimental): Disitamab Vedotin arm
  Interventions: Drug: Disitamab Vedotin Injection
- Paclitaxel (Experimental): Paclitaxel Arm
  Interventions: Drug: Paclitaxel Injection

INTERVENTIONS:
Drug: Disitamab Vedotin Injection — Phase II and III study ：2.5mg/kg, intravenous infusion，D1, every 2 weeks
  Other Names: DV,RC48
  Arms: Disitamab Vedotin; Disitamab Vedotin + Cadonilimab
Drug: Cadonilimab Injection — Phase II and III study ：6.0mg/kg, intravenous infusion，D1, every 2 weeks.
  Other Names: AK104, Cadonilimab Injection
  Arms: Disitamab Vedotin + Cadonilimab
Drug: Paclitaxel Injection — Phase II and III study ：Calculate dosage based on body surface are,160mg/m2,intravenous infusion，D1,D8 every 3 weeks
  Arms: Paclitaxel

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of Disitamab Vedotin Combined with Cadonilimab in subjects with HER2-expressing locally advanced or metastatic gastric cancer and gastroesophageal junction adenocarcinoma after progression on first-line therapy.

DETAILED DESCRIPTION:
This is an open-label, randomized, multicenter, Phase II/III Study designed to evaluate safety and efficacy of Disitamab Vedotin Combined with Cadonilimab in subjects with HER2-expressing locally advanced or metastatic gastric cancer and gastroesophageal junction adenocarcinoma after progression on first-line therapy.

This clinical study was divided into two parts, phase II and III.Part I: Phase II study primary objectives of the study are to evaluate the efficacy and safety of Disitamab Vedotin Combined with Cadonilimab versus Disitamab Vedotin versus paclitaxel in subjects with HER2-expressing locally advanced or metastatic gastric cancer and gastroesophageal junction adenocarcinoma after progression on first-line therapy.

Part II: Phase III study primary objectives of the study are to evaluate the efficacy and safety of Disitamab Vedotin Combined with Cadonilimab versus paclitaxel in subjects with HER2-expressing locally advanced or metastatic gastric cancer and gastroesophageal junction adenocarcinoma after progression on first-line therapy.

Tumor assessments, including radiological assessments by CT/MRI scans will be performed at Screening and subsequently every 6 weeks (±7 days) until disease progression, death, the start of new anticancer therapy, or patient's withdrawal of consent (whichever occurs first).

All patients who discontinue treatment will be followed for survival every 3 months until death, lost to follow-up, withdrawal of consent for survival follow-up, or end of study (whichever comes first).

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily agreed to participate in the study and signed an informed consent form;
2. Age 18-75 years(both 18 and 75);
3. Expected survival ≥ 12 weeks
4. ECOG physical condition score of 0 or 1
5. Locally advanced or metastatic gastric adenocarcinoma (including adenocarcinoma of the gastroesophageal junction) confirmed by histology and/or cytology
6. Subjects will only have failed or been intolerant to prior standard first-line therapy (excluding paclitaxel), with no restriction on prior treatment with a PD-1/PD-L1 inhibitor.
7. Confirmation of HER2 (IHC 1+, 2+, or 3+) and PD-L1 expression: for Phase II enrolled subjects, results of investigator-confirmed HER2 and PD-L1 expression will be accepted; for Phase III enrolled subjects, HER2 and PD-L1 expression will be accepted only as results from the central laboratory.
8. Bone marrow function:

   1. Hemoglobin ≥ 9 g/dL (no blood transfusion and no erythropoietin treatment within 2 weeks prior to the examination);
   2. Absolute neutrophil count ≥ 1.5 × 109/L (must not receive granulocyte colony-stimulating factor treatment within 2 weeks prior to the examination)
   3. Platelet count ≥ 90 × 109/L (no platelet transfusion or treatment with recombinant human thrombopoietin within 2 weeks before the test);
9. Liver function (based on normal values at the Clinical Trials Center):

   1. Serum total bilirubin ≤ 1.5 times the upper limit of normal (ULN);
   2. Alanine aminotransferase (ALT) and Mentholatum aminotransferase (AST) ≤ 2.5 × ULN in the absence of hepatic metastases; ALT and AST ≤ 5 × ULN in the presence of hepatic metastases;
10. Renal function (based on normal values at the Clinical Trials Center):

    Blood creatinine ≤ 1.5 x ULN, or creatinine clearance (CrCl) ≥ 60 mL/min calculated by the Cockcroft-Gault formula method, or measured 24-hour urine CrCl ≥ 60 mL/min;
11. Coagulation:

    1. Prothrombin time (PT) ≤ 1.5 x ULN;
    2. Thrombin time (TT) ≤ 1.5 × ULN;
    3. Activated partial thromboplastin time (APTT) ≤ 1.5×ULN;
12. Cardiac function:

    * New York Heart Association (NYHA) classification <3;
    * Left ventricular ejection fraction (LVEF) ≥ 50%;
13. The subject is able to provide specimens for central laboratory testing/review (at least 5 tissue sections) from the site of the primary or metastatic focus of the tumor within 3 years, preferably specimens taken after failure of first-line therapy;
14. Have at least one measurable lesion according to RECISTv1.1 criteria;
15. For female subjects: should be surgically sterilized, post-menopausal, or agree to use a medically approved contraceptive method (e.g., IUD, birth control pills, or condoms) for the duration of the study treatment and for 6 months after the end of the study treatment period; must have had a negative blood pregnancy test within 7 days prior to the study drug administration and must not be breastfeeding; and must not donate eggs for a period of 6 months from the time of signing of the informed consent form to the time of the last administration of the study drug. No egg donation for 6 months. For male subjects: should be surgically sterilized or agree to use a medically approved method of contraception during and for 6 months after the end of study treatment; no sperm donation from the time of signing the informed consent until at least 4 months after the last dose of study drug;
16. Be able to understand the requirements of the trial and be willing and able to comply with the trial and follow-up procedures.

Exclusion Criteria:

1. Metastatic CNS and/or meningeal carcinomatosis；
2. prior treatment with any antibody-drug conjugate including Disitamab Vedotin For Injection; prior treatment with cardinolizumab
3. Prior anti-cancer therapy resulting in toxicity that has not recovered to CTCAE (version 5.0) ≤ Grade 1 (except for hair loss, hyperpigmentation, or other conditions that do not increase the risk of the subject's use of the drug determined by the investigators;
4. Radical radiotherapy within 3 months prior to study dosing; palliative radiotherapy 2 weeks prior to dosing is permitted, at a dose that meets local diagnostic criteria for palliative care and with radiotherapy coverage of less than 30% of the bone marrow area;
5. Prior major surgery within 4 weeks before study dose start and incomplete recovery
6. Received a live vaccine within 28 days prior to the start of the first study dose or plan to receive any vaccine during the study period
7. Third interstitial effusion associated with clinical symptoms or that requires symptomatic treatment;
8. Ongoing grade ≥2 sensorimotor or motoneuropathy;
9. serum virology (based on site normal values):

   1. Positive Hepatitis B virus surface antigen (HBsAg) test result with a positive HBV DNA copy number;
   2. Positive test result for Hepatitis C Antibody (HCVAb) (enrollment in the study is only possible if the PCR test result for HCV RNA is negative);
   3. Positive test result for human immunodeficiency virus antibody (HIVAb).；
10. Serious arterial/venous or cardiovascular accidents, such as deep vein thrombosis ( except asymptomatic interstitial vein thrombosis which does not require special treatment), pulmonary embolism, cerebral infarction, cerebral hemorrhage, myocardial infarction, angina pectoris, etc., except for lacunar cerebral infarction, which is asymptomatic and does not require clinical intervention, have occurred in the last 6 months prior to the study drug administration;
11. Tumor lesions with bleeding tendency (e.g., presence of active ulcerated tumor lesions with a positive fecal occult blood test, history of vomiting blood or black stools within 2 months prior to signing the informed consent form, risk of gastrointestinal hemorrhage in the judgment of the investigator, etc.), or receipt of blood transfusion 4 weeks prior to study drug administration;;
12. The occurrence of an active or progressive infection requiring systemic treatment (trial drug may be initiated 2 weeks after completion of anti-infective therapy);
13. The presence of unsteady controlled systemic disease as judged by the investigator, including diabetes and hypertension, hepatocirrhosis, interstitial pneumonitis, and obstructive lung disease.
14. The existence of active autoimmune disease requiring systemic therapy (e.g., use of immunomodulatory agents, corticosteroids, or immunosuppressive agents) within 2 years prior to the start of study dosing, allowing for related replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for renal or pituitary insufficiency);
15. Other malignancy within 5 years prior to the start of study dosing, with the exception of the following: malignancies that are expected to resolve with treatment (including, but not limited to, adequately treated thyroid cancer, carcinoma in situ of the cervix, basal or squamous cell skin cancer, or ductal carcinoma in situ of the breast treated by radical surgery);
16. prior history of allogeneic hematopoietic stem cell transplantation or organ transplantation;
17. known hypersensitivity to immunosuppressants and any other antibody-drug conjugate and their components and any of the drugs in this study;
18. women who are pregnant or breast-feeding;
19. Any other disease, metabolic abnormality, physical examination abnormality, or laboratory test abnormality that, in the judgment of the Investigator, gives reason to suspect that the subject has a disease or condition that is unsuitable for the use of the study medication, would interfere with the interpretation of the results of the study, or puts the subject at a high risk of developing a condition;
20. subjects whose participation in this study is estimated to be insufficiently adherent or who, in the judgment of the investigator, have other factors that make them unsuitable for participation in this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-02-22 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Objective remission rate (ORR) (Phase II) | Up to approximately 2 years
  ORR assessed according to the evaluation criteria for the efficacy of solid tumors (RECIST 1.1)
Percentage of Participants With Adverse Events (AEs)(Phase II) | Up to approximately 2 years
  Number of participants with adverse effects of treatment. Frequency and severity of adverse effects of treatment as assessed by NCI CTCAE v5.0
Progression-Free Survival(PFS) （IRC）（ Phase III) | Up to approximately 2 years
  PFS was defined as the time from random assignment to the onset of disease progression (as assessed by the IRC according to RECIST v1.1 criteria) or death (whichever event occurs first)
Overall Survival (OS)(Phase III) | Up to approximately 2 years
  OS was defined as the time from the date of randomization to the date of death from any cause.

SECONDARY OUTCOMES:
Progression-Free Survival(PFS)（investigator）(Phase II and Phase III) | Up to approximately 2 years
  PFS was defined as the time from random assignment to the onset of disease progression (as assessed by the IRC according to RECIST v1.1 criteria) or death (whichever event occurs first)
Overall Survival (OS)(Phase II) | Up to approximately 2 years
  OS was defined as the time from the date of randomization to the date of death from any cause.
Objective remission rate (ORR) （investigator） (Phase III) | Up to approximately 2 years
  ORR assessed according to the evaluation criteria for the efficacy of solid tumors (RECIST 1.1)
Disease Control Rate (DCR) (Phase II and Phase III) | Until progression, assessed up to approximately 2 years
  Percentage of patients with complete response, partial response, or stable disease for a certain period of time according to RECIST v1.1.
Duration of response (DoR) (Phase II and Phase III) | Until progression, assessed up to approximately 2 years
  Defined as the time from the date of first documented response (CR/PR) until the first progression or death in the absence of disease progression by Investigators assessment according to RECIST 1.1
Type, incidence, relatedness, severity, and seriousness of AEs | Up to approximately 2 years
  According to NCI-CTCAE Version 5.0 per each treatment arm
Incidence of laboratory tests abnormalities | Up to follow-up period, approximately 2 years
  To be summarized using descriptive statistics
Incidence of ECG abnormalities | Up to follow-up period, approximately 2 years
  To be summarized using descriptive statistics
Incidence of echocardiograms abnormalities | Up to approximately 2 years
  Change from baseline of LVEF

CONTACTS AND LOCATIONS:
Overall Officials: Jianmin Fang, Ph.D, Study Director — RemeGen Co., Ltd.
Locations (12):
- China (12):
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - The First Affiliated Hospital of Xiamen University, Xiamen, Fujian
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjiang
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Hubei Cancer Hospital, Wuhan, Hubei
  - Hunan Cancer Hospital, Changsha, Hunan
  - Xuzhou Central Hospital, Xuzhou, Jiangsu
  - Shandong Cancer Hospital, Jinan, Shandong
  - The Affiliated Hospital of Qingdao University, Qingdao, Shandong
  - Ruijin Hospital Affiliated to Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality
  - West China Hospital of Sichuan University, Chengdu, Sichuan
  - Yunnan Cancer Hospital, Kunming, Yunnan